CLINICAL TRIAL: NCT01594463
Title: Third Trimester Routine Ultrasound in Low-risk Pregnancies : Comparison of Two Timing Periods Procedure for Screening Intrauterine Growth Restriction
Brief Title: Routine Ultrasound Screening in the Third Trimester
Acronym: RECRET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010/090/HP
Record Dates: First submitted 2012-04-27; First posted 2012-05-09 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Fetal Growth Retardation; High-Risk Pregnancy
Keywords: Intrauterine growth restriction; Screening; Ultrasound; Perinatal morbidity; Maternal complications
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- late ultrasound examination (Experimental): late examination between 34+1 weeks to 35+6 weeks.
  Interventions: Other: ultrasound examination
- early ultrasound examination (Experimental): early examination between 30+1 weeks to 31+6 weeks
  Interventions: Other: ultrasound examination

INTERVENTIONS:
Other: ultrasound examination — ultrasound examination between week 30+1 weeks to 31+6 weeks
  Arms: early ultrasound examination
Other: ultrasound examination — ultrasound examination between 34+1 weeks to 35+6 weeks
  Arms: late ultrasound examination

SUMMARY:
Late intrauterine growth restriction is infrequently diagnosed with an overall sensitivity of 40 % in low-risk pregnancies. In addition, late intrauterine growth restriction may be associated with intrauterine death and poor neonatal outcomes i.e. birth asphyxia and hospitalization in intensive care unit. The investigators hypothesis that a later third trimester routine ultrasound may be more accurate to diagnose late intrauterine growth restriction.

ELIGIBILITY:
Inclusion Criteria:

* Accurate gestational dating using crown-rump length at 11-14 weeks
* Singleton pregnancy
* Primiparity
* Normal First trimester (11-14 weeks) and second trimester (20-25 weeks) scans
* Maternal age > 18 years
* No maternal opposition for the study

Exclusion Criteria:

* Maternal diseases i.e. chronic renal disease, hypertension, diabetes, collagen vascular disease, antiphospholipid syndrome
* Pregnancies with congenital anomalies or foetal growth restriction diagnosed before 30 weeks of gestation

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3760 (Actual)
Dates: Start 2012-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number of small for gestational age infant screened by a routine ultrasound in the third trimester (sensitivity). | At birth
  SGA infant and intrauterine growth restriction are defined using a threshold below the tenth percentile for customized birth weight or customized estimated birth weight.

SECONDARY OUTCOMES:
Number of neonate with a customized birth weight upper the tenth percentile adequately screened by a routine ultrasound in the third trimester (specificity). | At birth
Number of prenatal consultations, ultrasound scans performed, maternal hospitalization, labor induction, and caesarean section induced by the third trimester routine ultrasound | After the delivery
Maternal complications and neonatal outcomes. | In the postpartum period

CONTACTS AND LOCATIONS:
Overall Officials: Eric VERSPYCK, Pr, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France